CLINICAL TRIAL: NCT02763605
Title: Retrospective Study of the in Vivo Confocal Microscopic Findings and the Treatment Outcome of Acanthamoebic Keratitis
Brief Title: Retrospective Study of Acanthamoebic Keratitis During the Past 10 Years
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201312046RINB
Record Dates: First submitted 2016-04-12; First posted 2016-05-05 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Acanthamoeba Keratitis
Keywords: Acanthamoeba Keratitis; in vivo confocal microscopic
MeSH Terms: conditions — Acanthamoeba Keratitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- patients diagnosed with acanthamoeba keratitis: Inclusion Criteria:
  - All patients presenting to National Taiwan University Department from Jun. 1st, 2003 to dec. 30th , 2016 with the tissue proven corneal AK will be included.
  Exclusion Criteria
  - Patients with tissue proven corneal AK during from Jun. 1st, 2003 to dec. 30th , 2016, but without in vivo confocal data, or complete chart records.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Acanthamoebic keratitis is an important corneal disease which may cause severe complication. The difficulty in diagnosis, the difficulty in treatment, and the long treatment process are factors leading to the poor prognosis of these patients. In this retrospective study, the investigators try to analyze the tissue proven Acanthamoebic keratitis diagnosed in our hospital. The investigators will focus on the in vivo confocal microscopic results, the medical history and the medical/surgical treatment outcome. The investigators will collect the tissue proven cases according to the data provided by laboratory diagnosis department and pathological department. The in vivo confocal microscopic results will be collected and analyzed. The investigators will also look through the photography of the external eyes from data stored in PAC system. The medical history and treatment outcome will be studied from clinical chart review. From this study, the investigators aimed to find out a easy way of diagnosing Acanthamoebic keratitis from in vivo confocal microscopy, and find out a better way for treatment.

DETAILED DESCRIPTION:
Acanthamoeba keratitis (AK), caused by a pathogenic amoeba, is a sight-threatening corneal infection with severe pain, epithelial defect, epithelial haze, pseudodendrites, and, most characteristically, radial keratoneuritis. The corneal infection of AK was first recognized in the mid 1970s. Since then, a growing number of AK cases were diagnosed, mainly resulting from improper use of soft contact lenses.

Clinical diagnosis of AL is difficult, especially in the early phases of the disease, and it often is misdiagnosed and treated as a herpes simplex infection. It was reported a diagnostic delay of more than 18 days between onset of symptoms and start of anti- amoebic treatment results in a poor disease progress. While definitive diagnosis is made by confirmation of Acanthamoeba cysts or trophozoites in corneal lesions by staining, corneal biopsy, or tissue culturing.

In vivo confocal microscopy was considered useful in the rapid diagnosis of AK. The Acanthamoeba cysts were observed almost exclusively in the epithelial cell layer as highly reflective, round or stellate, high-contrast particles with a diameter of 10 to 20 μm. It was suggested that invasion of Acanthamoeba cysts into Bowman's layer may be a useful predictor for a persistent clinical course. The trophozoites are pear-shaped or irregularly wedge-shaped structures, some surrounded by a brilliant halo some exhibiting fine pseudopodia-like extensions, with mean size of 30.2 µm (range 19.2-55.6μm). It was reported to present in cornea stroma. Highly reflective activated keratocytes forming a honeycomb pattern change was reported to be present around the keratoneuritis. In addition, infiltration of inflammatory cells, possibly polymorphonuclear cells, was observed along with the keratocytes in cases of AK. However, the in vivo confocal microscopic findings in patients with AK is still limited. Some clinical findings may not be correlated with the reports published before.

John K.G. et al recommended clinical treatment toward Acanthamoeba keratitis using Diamidine and Biguanide which are the only two proofed Acanthamoeba cysticidal medication, while Metronidazole is effective in vivo but not in vitro. Topical steroid was considered rather controversial but important and beneficial. It was recommended to use a minimum of 2 weeks of Biguanide prior to the use of topical steroid for inflammation control. When Acanthamoeba keratitis was diagnosed early in the disease course, topical steroid can be spared for the immediate using Diamidine and Biguanide to kill pathogen. In a United Kingdom multicenter study of 218 patients, the average duration of medical therapy was 6 months (range, 0.5 to 29 months). In 2011, a little over half of respondents using corticosteroids in the treatment of Acanthamoeba keratitis. Surgical managements including epithelial debridement, cryotherapy and corneal graft surgery may itself be therapeutic if performed early and promote penetration. Therefore, when Acanthamoeba keratitis was suspected, a long-term and immediate medical treatment may be needed ,and the use of topical steroid toward Acanthamoeba keratitis is still worth investigating.

ELIGIBILITY:
Inclusion Criteria:

* presenting to National Taiwan University Department from Jun. 1st, 2003 to dec. 30th , 2016
* suspecting Acanthamoeba Keratitis by the ophthalmologist
* drug treatment as Acanthamoeba Keratitis successed
* tissue proved to be Acanthamoeba Keratitis
* referred from the other hospital with the diagnose of Acanthamoeba Keratitis

Exclusion Criteria

* patients suspect corneal Acanthamoeba Keratitis from Jun. 1st, 2003 to dec. 30th , 2013, but without in vivo confocal data, or complete chart records.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The in vivo confocal microscopic data and medical records of all recruited patients diagnosed with Acanthamoeba Keratitis will be reviewed after approved by the NTUH Institutional Review Board Committee. Data collected include patient demographics (age, gender), local findings, external eye photos, treatment course and treatment outcome. In vivo confocal microscope exam results will be compared with the clinical manifestation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with typical image finding under an in vivo confocal microscope (Confoscan 3.4.1; Nidek Technologies, Padova, Italy) | through study completion, an average of about 10 year microscope diagnosis and disease progress prediction of patients with Acanthamoe

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, MD,PHD, Study Director — professor of National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Naginton J, Watson PG, Playfair TJ, McGill J, Jones BR, Steele AD. Amoebic infection of the eye. Lancet. 1974 Dec 28;2(7896):1537-40. doi: 10.1016/s0140-6736(74)90285-2. No abstract available. PMID 4140981
- [Background] Mathers WD, Sutphin JE, Folberg R, Meier PA, Wenzel RP, Elgin RG. Outbreak of keratitis presumed to be caused by Acanthamoeba. Am J Ophthalmol. 1996 Feb;121(2):129-42. doi: 10.1016/s0002-9394(14)70577-x. PMID 8623882
- [Background] Claerhout I, Goegebuer A, Van Den Broecke C, Kestelyn P. Delay in diagnosis and outcome of Acanthamoeba keratitis. Graefes Arch Clin Exp Ophthalmol. 2004 Aug;242(8):648-53. doi: 10.1007/s00417-003-0805-7. PMID 15221303
- [Background] Winchester K, Mathers WD, Sutphin JE, Daley TE. Diagnosis of Acanthamoeba keratitis in vivo with confocal microscopy. Cornea. 1995 Jan;14(1):10-7. PMID 7712728
- [Background] Matsumoto Y, Dogru M, Sato EA, Katono Y, Uchino Y, Shimmura S, Tsubota K. The application of in vivo confocal scanning laser microscopy in the management of Acanthamoeba keratitis. Mol Vis. 2007 Jul 25;13:1319-26. PMID 17679934
- [Background] Parmar DN, Awwad ST, Petroll WM, Bowman RW, McCulley JP, Cavanagh HD. Tandem scanning confocal corneal microscopy in the diagnosis of suspected acanthamoeba keratitis. Ophthalmology. 2006 Apr;113(4):538-47. doi: 10.1016/j.ophtha.2005.12.022. PMID 16581415
- [Background] Yokogawa H, Kobayashi A, Yamazaki N, Ishibashi Y, Oikawa Y, Tokoro M, Sugiyama K. Bowman's layer encystment in cases of persistent Acanthamoeba keratitis. Clin Ophthalmol. 2012;6:1245-51. doi: 10.2147/OPTH.S34695. Epub 2012 Aug 2. PMID 22927735
- [Background] Rezaei Kanavi M, Naghshgar N, Javadi MA, Sadat Hashemi M. Various confocal scan features of cysts and trophozoites in cases with Acanthamoeba keratitis. Eur J Ophthalmol. 2012;22 Suppl 7:S46-50. doi: 10.5301/ejo.5000139. PMID 22427148
- [Background] Pfister DR, Cameron JD, Krachmer JH, Holland EJ. Confocal microscopy findings of Acanthamoeba keratitis. Am J Ophthalmol. 1996 Feb;121(2):119-28. doi: 10.1016/s0002-9394(14)70576-8. PMID 8623881
- [Background] Shiraishi A, Uno T, Oka N, Hara Y, Yamaguchi M, Ohashi Y. In vivo and in vitro laser confocal microscopy to diagnose acanthamoeba keratitis. Cornea. 2010 Aug;29(8):861-5. doi: 10.1097/ICO.0b013e3181ca36b6. PMID 20508505
- [Background] Dart JK, Saw VP, Kilvington S. Acanthamoeba keratitis: diagnosis and treatment update 2009. Am J Ophthalmol. 2009 Oct;148(4):487-499.e2. doi: 10.1016/j.ajo.2009.06.009. Epub 2009 Aug 5. PMID 19660733
- [Background] Radford CF, Lehmann OJ, Dart JK. Acanthamoeba keratitis: multicentre survey in England 1992-6. National Acanthamoeba Keratitis Study Group. Br J Ophthalmol. 1998 Dec;82(12):1387-92. doi: 10.1136/bjo.82.12.1387. PMID 9930269
- [Background] Oldenburg CE, Acharya NR, Tu EY, Zegans ME, Mannis MJ, Gaynor BD, Whitcher JP, Lietman TM, Keenan JD. Practice patterns and opinions in the treatment of acanthamoeba keratitis. Cornea. 2011 Dec;30(12):1363-8. doi: 10.1097/ICO.0b013e31820f7763. PMID 21993459